CLINICAL TRIAL: NCT07337759
Title: Placental Weight and Surface as an Indicator of Placental Insufficiency and Adverse Perinatal Outcomes
Brief Title: Fetus Programming and Long Active Outcomes, Interaction Between Mother, Placenta and Fetus in Perinatal and Methabolic Disbalansces-focusing Diabetic Pregnancies
Status: Completed | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Miroslava Gojnic Dugalic, Prof. dr, University of Belgrade
Other Study IDs: 1880/6
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Placental Insufficiency Hypertensive Disorders of Pregnancy Diabetes Mellitus in Pregnancy Thrombophilia in Pregnancy Adverse Perinatal Outcomes
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Appropriate-for-Gestational-Age Placenta (AGA-P): regnant women whose placentas had a weight between the 10th and 90th percentile for gestational age.
  Interventions: Other: No intervention (observational study)
- Small-for-Gestational-Age Placenta (SGA-P): Pregnant women whose placentas had a weight below the 10th percentile for gestational age.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — observational study

SUMMARY:
The placenta is a temporary but essential organ that develops during pregnancy and supports the growth and survival of the fetus. It delivers oxygen and nutrients from the mother to the baby and removes waste products from the fetal circulation. Proper placental development and function are critical for a healthy pregnancy and good outcomes for both the mother and the newborn.

When the placenta does not grow or function properly, this condition is known as placental insufficiency. Placental insufficiency may lead to serious pregnancy complications, such as poor fetal growth, preterm birth, low birth weight, low Apgar scores, and increased risk of illness or death around the time of birth. In some cases, placental dysfunction may also contribute to maternal complications, including pregnancy-related hypertension.

Previous research has shown that simple physical characteristics of the placenta-such as its weight, size, thickness, and surface area-may reflect how well the placenta functions. Placentas that are smaller than expected for a given gestational age may indicate long-standing problems with blood flow between the mother and the fetus. However, these measurements are not yet routinely used as clinical markers of risk.

The purpose of this study was to examine whether placental weight, placental surface area, placental disk weight, and related histopathological changes are associated with adverse perinatal outcomes. The study included both healthy pregnant women and women with medical conditions known to affect pregnancy, such as hypertension, diabetes mellitus, and thrombophilia. Special attention was given to placentas classified as small for gestational age (SGA-P) compared with placentas appropriate for gestational age (AGA-P).

ELIGIBILITY:
Inclusion Criteria: Pregnant women who delivered at the Clinic of Gynecology and Obstetrics, University Clinical Centre of Serbia

* Singleton pregnancy
* Available placental examination after delivery
* Available clinical and perinatal outcome data
* Gestational age at delivery ≥24 weeks

Exclusion Criteria:

Multiple pregnancy (e.g., twins or higher-order gestations)

* Major congenital or chromosomal fetal anomalies
* Intrauterine fetal demise
* Conditions directly affecting placental weight (e.g., placental mosaicism)
* Incomplete clinical, placental, or histopathological data

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with singleton pregnancies who delivered at the Clinic of Gynecology and Obstetrics, University Clinical Centre of Serbia. The study population includes both healthy pregnant women and women with maternal comorbidities such as hypertensive disorders, diabetes mellitus, and thrombophilia. Placentas were examined after delivery and classified according to placental weight for gestational age.
Sampling Method: Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-01-04 (Actual); Study Completion 2026-01-04 (Actual)

PRIMARY OUTCOMES:
Adverse perinatal outcome defined as at least one of the following: delivery before 34 gestational weeks, birth weight below 2200 g, or Apgar score <7 at 5 minutes. | From delivery to 5 minutes after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of Gynecology and Obstetrics, University Clinical Center of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No